CLINICAL TRIAL: NCT06332521
Title: Infant Crying, a Bioacoustic Prognostic Signal for Neurodevelopment
Acronym: BABYCRY_1000
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 23CH296; ANSM (Other: 2024-A00286-41)
Record Dates: First submitted 2024-03-20; First posted 2024-03-27 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Newborn; Vitality; Premature Infants; Infant Development
Keywords: Newborn; Crying
MeSH Terms: conditions — Premature Birth; Crying

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- birth of term babies: Study of crying in a group of newborns (birth of term babies)
  Interventions: Other: Acoustic signal analysis method
- Premature babies: Study of crying in a group of newborns (Premature babies )
  Interventions: Other: Acoustic signal analysis method

INTERVENTIONS:
Other: Acoustic signal analysis method — Evaluate at birth in 2 characterized populations of babies born at term or prematurely, the correlation between bioacoustic characteristic of a cry specific to each baby, with the neurodevelopmental data at 2 years.

SUMMARY:
Crying is a vital communication signal for the baby. Product of a complex physiological process, it reflects not only the organization and functioning of the cortical central nervous system and the function of sympathetic and parasympathetic autonomic regulation but also the integrity of three entities: the lungs responsible for ventilatory mechanics and respiratory rhythm, the larynx and its vocal cords as a phonatory organ, and the oropharyngeal tract guaranteeing the resonance of the sound emitted by the vocal cords.

Crying is usually caused by pain, discomfort, hunger, or separation from parents or other caregivers. Crying carries essential information from birth, the expression of which depends closely on the neuroanatomical and functional brain integrity of the child. On a bioacoustic level, crying consists of sequences of complex acoustic signals produced by the vocal folds and filtered by the vocal tract. The vibration frequency of the vocal cords determines the cry's fundamental frequency f0 (and the harmonic frequencies), which is responsible for its more or less low or high pitch. Other acoustic cues also characterize each baby's cry.

DETAILED DESCRIPTION:
The objective of the Baby's cry 1000/100 study is to evaluate the acoustic characteristics of crying at birth, of term and premature babies and to correlate them with neurodevelopmental outcomes at 2 years of age to see if the bioacoustic characteristics of crying at birth could be predictive of the baby's neurofunctional integrity.

To achieve this objective, the investigators wish to document a large bank of recordings of the crying of term or premature babies by relying on deep learning and artificial intelligence approaches, making it possible to process large databases quickly, evaluate the links between acoustics of crying and clinical data at the birth of full-term babies who will benefit from systematic neurodevelopmental monitoring at 2 years (Bayley scale).

ELIGIBILITY:
Inclusion Criteria:

* For a full-term baby > 37 weeks
* For a premature baby < 37 weeks
* Born in the maternity ward of the Saint-Etienne University Hospital
* Holder of parental authority having received informed information about the study and their right to object
* Holder of parental authority affiliated to or beneficiary of a social security system
* Eutrophic between the 10th and 90th percentile on the neonatal curves)

Exclusion Criteria:

* Refusal of participation by the holder of parental authority
* Antenatal pathology, nor perinatal asphyxia
* Holder of minor parental authority
* Holder of parental authority under curatorship or guardianship
* Abnormal T1 audiological screening test.

Max Age: 4 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Full-term baby > 37 weeks Premature baby < 37 weeks
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Fundamental frequency f0 (Hz) | At inclusion
  Fundamental frequency f0 (Hz) defined from a crying sequence, the most characteristic elementary index of their individual bioacoustic signature.
Bailey-4 quantitative scale | At 2 years
  neurodevelopment at age 2 measured by the Bailey-4 quantitative scale. The final score is from 40 (Very weak neurodevelopment) to 160 (Very good neurodevelopment)

SECONDARY OUTCOMES:
Percentage voiced frames | At inclusion
  Other bioacoustic characteristics measurable in each bioacoustic sequence
Harmonics of f0 (Hz) | At inclusion
  Other bioacoustic characteristics measurable in each bioacoustic sequence : vibration frequency of the vocal cords, defining a +/- low or high tone
Median pitch f0 (Hz) | At inclusion
  Other bioacoustic characteristics measurable in each bioacoustic sequence
Harmonicity (dB) | At inclusion
  Other bioacoustic characteristics measurable in each bioacoustic sequence
Jitter (Percentage), | At inclusion
  Other bioacoustic characteristics measurable in each bioacoustic sequence
Q25 (Percentage) | At inclusion
  Other bioacoustic characteristics measurable in each bioacoustic sequence : rapid amplitude fluctuations occurring at frequencies between 30 and 150 Hz
Median Cepstral Peak Prominence (CPP) (dB) | At inclusion
  The CPP makes it possible to quantify the "quality" of the voice and the acoustic signal and its degree of harmonicity as opposed to the severity of the dysphonia

CONTACTS AND LOCATIONS:
Overall Officials: HUGUES PATURAL, MD-PhD, Principal Investigator — CHU DE SAINT-ETIENNE; Nicolas MATHEVON, PhD, Study Chair — Saint-Etienne University
Locations (1):
- Chu de Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No